CLINICAL TRIAL: NCT03838315
Title: Effects of Neural Mobilization With or Without Soft Tissue Mobilization in Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Noor Abid, Research Associate, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIRS-IUISB/MphilOPT/002
Record Dates: First submitted 2019-02-09; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy,; Neural Mobilizations,; Soft Tissue Mobilization
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Intervention Model Description: Subjects will be assigned randomly into two groups: Neural Mobilization with Soft tissue mobilization and Neural mobilization without Soft tissue mobilization.A coin will be flipped at start of data collection for the first patient to be assigned odd number and included in Neural mobilization with Soft tissue mobilization group. Later on odd and even numbered subjects will be included in specific group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilization with Soft Tissue Mobilization (Experimental): Neural Mobilization with Soft Tissue Mobilization group will be assessed by spurling's test and than will involved in treatment protocol i.e Cervical Traction, Hot packs, Neural mobilization Techniques which involve Median, Radial and Ulnar Nerve Mobilization and Post Isometric Relaxation Techniques.
  Frequency for Neural mobilization is 3 sets of 10 repetitions for each and duration of 15minute. Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 40mints each session)
  Interventions: Other: Neural Mobilization with Soft Tissue Mobilization
- Neural mobilization without Soft Tissue Mobilization (Active Comparator): Neural Mobilization without Soft Tissue Mobilization group will be assessed by spurling's test and than will involved in treatment protocol i.e Cervical Traction, Hot packs, Neural Mobilization Participant will be scheduled to attend 12 treatment session (3 sessions every week for 4 weeks, 30mints each session)
  Interventions: Other: Neural Mobilization without Soft Tissue Mobilization

INTERVENTIONS:
Other: Neural Mobilization with Soft Tissue Mobilization — Cervical Traction for 10mints 7%of body weight with 7 second hold time and 5 second rest time.
  Hot Pack for 10mints. Neural mobilization technique includes Median, Radial and Ulnar nerve mobilization. Frequency for neural mobilization is 3 sets of 10 repetitions for each and duration of 10minute.
  •Post isometric relaxation technique
  Arms: Neural Mobilization with Soft Tissue Mobilization
Other: Neural Mobilization without Soft Tissue Mobilization — Cervical Traction for 10mints 7%of body weight with 7 second hold time and 5 second rest time.
  * Hot Pack
  * Neural mobilization technique includes Median, Radial and Ulnar nerve mobilization Frequency for neural mobilization is 3 sets of 10 repetitions for each and duration of 10minute.
  Arms: Neural mobilization without Soft Tissue Mobilization

SUMMARY:
This study will evaluate Effects of Neural Mobilization with or without Soft Tissue Mobilization in Cervical Radiculopathy, half of the subjects will receive treatment of Neural Mobilization along with Soft Tissue Mobilization whereas half of the subjects will receive only Neural Mobilization.

DETAILED DESCRIPTION:
Neural mobilization and Soft Tissue Mobilization both treatments are used to treat Cervical Radiculopathy but they work differently.

Neural mobilization technique is different for all 3 nerves i.e Radial, ulnar and median. Neural Mobilization Technique target the single nerve which is being compressed and showing symptoms.

Soft Tissue Mobilization include traction which decompresses the nerve and stretches the surrounding muscles along with help to reduce pain and tingling sensation. whereas hot pack helps to increase blood circulation and warm up muscles and isometric exercises provide strengthening and build endurance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age 18 to 55years
* Patients having pain more than 3months
* Radiating pain in one of the upper limb
* Spurling's test positive

Exclusion Criteria:

* Traumatic injury of upper limb or cervical spine
* Vertebral artery test positive(dizziness, vomiting, diplopia, drop attacks etc)
* Patient asymptomatic for pain but symptomatic for tingling and paraesthesia
* Circulatory disturbance of upper extremity
* Known history of high level of spinal cord injury and malignancy
* Thoracic Outlet syndrome

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-05-20 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Neck Pain Numeric Scale | 4weeks
  Pain intensity in one of the upper limb is measured by Numeric pain scale in which "0"

SECONDARY OUTCOMES:
Neck Disability Index | 4weeks
  Neck disability index scale used to measure ability to manage neck pain in everyday life in terms of: Pain intensity, Personal care, Lifting, Reading, Headaches, and Concentration. In which "0" shows disability and "5" shows normal.